CLINICAL TRIAL: NCT04883723
Title: The Effect of Use of Manual Pressure and Shotblocker on Pain and Injection Satisfaction in the Application of Intramuscular Injection to the Ventrogluteal Region in Adult Patients
Brief Title: Effect of Manual Pressure and Shotblocker on Pain and Injection Satisfaction in Intramuscular Injection Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ali Kaplan, lecturer, TC Erciyes University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: Ali KAPLAN-Erciyes University
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Intramuscular Injection
Keywords: shotblocker; manual pressure; İntramuscular injection; pain; injection satisfaction
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: During the data collection, 120 individuals who met the inclusion criteria and were selected with the randomization list created on the computer constituted the sample of the study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experiment I (Shotblocker) Group (Experimental): Before the injection, the heart rate and blood pressure values of the patient were measured and recorded. The patient was placed in a prone position. The determined injection site was cleaned with a cotton pad with alcohol, with circular movements of 5 cm diameter from inside to outside, and the alcohol was allowed to dry. The protruding surface of the Shotblocker was placed in the area just before the injection, so that the needle entry point would not be contaminated. It was lightly pressed into the shotblocker with fingertips and the injection was performed. ShotBlocker has been removed after removing the needle. Visual comparison scale and injection satisfaction evaluation scale were applied to the patient in the first minute after the intramuscular injection. The obtained scores were recorded in the patient identification form. Pulse and blood pressure values were measured and recorded again. Finally, the patient introduction form was filled.
  Interventions: Device: Shotblocker
- Experiment II (Manual Pressure) Group (Experimental): Before the injection, the heart rate and blood pressure values of the patient were measured and recorded. The patient was placed in a prone position and the appropriate left or right ventrogluteal region was determined. Pressure was applied to the determined injection area with the thumb of the active hand for 10 seconds. Immediately after the application of pressure was terminated, the injection site was cleaned with an alcohol cotton pad with circular movements of 5 cm diameter from inside to outside and the alcohol was allowed to dry. With a single movement at a 90 ° angle, the compression area was entered quickly and the injection was performed. Visual comparison scale and injection satisfaction evaluation scale were applied to the patient in the first minute after the intramuscular injection. The obtained scores were recorded in the patient identification form. Pulse and blood pressure values were measured and recorded again. Finally, the patient introduction form was filled.
  Interventions: Other: Manual Pressure
- Control Group (No Intervention): The patients in the Manual Pressure group were given detailed information about the procedure and the research, and the patients who agreed to participate in the study were signed by an informed consent form. Before the injection, the heart rate and blood pressure values of the patient were measured and recorded. The patient was placed in a prone position and the appropriate left or right ventrogluteal region was determined. Injection was given using the normal intramuscular injection procedure. Visual comparison scale and injection satisfaction evaluation scale were applied to the patient in the first minute after the intramuscular injection. The obtained scores were recorded in the patient identification form. Pulse and blood pressure values were measured and recorded again. Finally, the patient introduction form was filled.

INTERVENTIONS:
Device: Shotblocker — Shotblocker is a small, flat, horseshoe-shaped plastic tool that can be used to reduce pain due to intramuscular injection, suitable for all age groups, without drug properties. It is used by keeping it on the skin surface during injection and has no side effects. Shotblocker has short, non-pointed blunt protrusions on one side that connect with the skin, there is a hole in the middle of the vehicle to expose the injection site. The protruding surface of the vehicle is placed in the area to be applied just before injection. The protrusions on the surface of the Shotblocker do not pierce the skin and provide a warning for the Door Control Theory, which is thought to exist regarding pain
  Arms: Experiment I (Shotblocker) Group
Other: Manual Pressure — The patient was placed in a prone position and the appropriate left or right ventrogluteal region was determined. Pressure was applied to the determined injection area with the thumb of the active hand for 10 seconds. Immediately after the application of pressure was terminated, the injection site was cleaned with an alcohol cotton pad with circular movements of 5 cm diameter from inside to outside, and the alcohol was allowed to dry. With a single movement at a 90 ° angle, the compression area was entered quickly and the injection was performed. Manual pressure reduces pain within the framework of the gate control theory. According to the gate control theory, when pressure is applied to an area, a fiber transmits the feeling of pressure instead of pain and ultimately the pain sensation is alleviated. There are many studies in the literature that prove the effectiveness of this method.
  Arms: Experiment II (Manual Pressure) Group

SUMMARY:
This study was planned as a single blind randomized controlled experimental study to investigate the effect of manual pressure applied before injection and ShotBlocker's pain and injection satisfaction due to intramuscular injection. The sample of the study consisted of a total of 120 patients over the age of 18 who applied to the Emergency Service of a public hospital and were requested Diclofenac Sodium 75mg / 3ml. The patients were included in the experiment I (shotblocker), experiment II (manual compression) and the control group with the randomization list created on the computer.

In the ShotBlocker group, the ShotBlocker was kept throughout the injection, and in the manual compression group, manual pressure was applied to the injection area for 10 seconds before injection, and in the control group, IM injection was applied without using any tools. Before the injection, the heart rate and blood pressure values of the patient were measured and recorded. Visual Comparison Scale and Injection Satisfaction Scale were administered to the patient in the first minute after the injection. Pulse and blood pressure values were measured and recorded again. Finally, the patient introduction form was filled. Parametric or nonparametric statistical tests and correlation test were used in the analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

* He has not had an IM injection in the last week,
* Upper respiratory tract infection patients in the Examination Department, where green field patients of the Emergency Service are located,
* Over the age of 18,
* No complications related to IM injections such as pain at the IM injection site, abscess, infection, tissue necrosis, hematoma,
* Does not have pain anywhere in the body that will affect the work result,
* Are conscious and have no communication problem,
* No vision or hearing problems,
* Not taking analgesic in the last 24 hours,
* Does not have any known chronic disease,
* No psychiatric disorder,
* Diclofenac sodium ampoule has been ordered,
* Can evaluate "Visual Comparison Scale and Injection Satisfaction Scale" correctly,
* Individuals who volunteered to participate in the study and signed the written informed consent form were included.

Exclusion Criteria:

* Not wanting to participate in the study,
* Patients who did not meet the study acceptance criteria were not included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-08-23 (Actual)

PRIMARY OUTCOMES:
Visual Benchmark Scale | Immediately after the injection
  It is a one-dimensional scale used in the measurement of pain. It was found that the sensitivity of the visual comparison scale was higher than other methods in the assessment of pain severity. The scale consists of a 100 mm long line. On one end there are the words "No Pain" and "Unbearable Pain" on the other. The patient is instructed to mark a point on the line that accurately reflects his or her pain. Between the onset of no pain and this point marked by the patient, it is measured and recorded.
Injection Satisfaction Rating Scale | Immediately after the injection
  The satisfaction level of the patients after injection was evaluated using a scale consisting of a 100 mm vertical line with "Very Satisfied" on one end and "Not Satisfied" on the other.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol